CLINICAL TRIAL: NCT00847600
Title: Pregnenolone Augmentation in the Treatment of Patients With Recent-Onset Schizophrenia: an 8-week, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Pregnenolone Augmentation in the Treatment of Patients With Recent-Onset Schizophrenia
Acronym: PREG-2008
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Technion and Shaar Menashe MHC, Technion and Shaar Menashe MHC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEN-8-11-08; 08TGF-1189 Stanley grant
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorders
Keywords: Schizophrenia; Neurosteroids; Pregnenolone; Augmentation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Pregnenolone (Experimental): 50 mg/day
  Interventions: Dietary Supplement: Pregnenolone
- 2 Placebo (Placebo Comparator): 1 caps.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pregnenolone — 50 mg, caps.
  Arms: 1 Pregnenolone
Dietary Supplement: Placebo — caps
  Arms: 2 Placebo

SUMMARY:
Pregnenolone (PREG) is a neurosteroid, which displays multiple effects on the central nervous system, and may be beneficial in the treatment of patients with schizophrenia. Our recent 8-week, randomized, double-blind trial among patients with chronic schizophrenia and schizoaffective disorders, in which PREG versus placebo and DHEA have been added to conventional or atypical antipsychotics have yielded encouraging results with low-dose PREG (30 mg/day; ClinicalTrials.gov identifier NCT00140192; Ritsner et al., in press). The goal of the present study is to evaluate the potential role of PREG's augmentation compared to placebo in the treatment of young patients with newly diagnosed schizophrenia or schizophreniform or schizoaffective disorders.

In a 8-week, randomized, double-blind placebo-controlled trial PREG (50 mg/day) or placebo capsules will be added to the stable ongoing antipsychotic treatment of 60 patients with recent-onset schizophrenia or schizophreniform or schizoaffective disorders. Participants will be assessed at baseline and after 2, 4, 6 and 8 weeks of treatment. A battery of research instruments will be used for assessment of psychopathology, cognitive functions, side effects, general functioning and quality of life. In addition blood PREG levels will be monitored at baseline and during the study. The study is powered to detect moderate between-group effects on persistent positive, negative and cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18-40 years of age, any ethnic group, either sex.
2. DSM-IV criteria for schizophrenia, schizophreniform or schizoaffective disorders (36).
3. Duration of illness less than 5 years since onset first psychotic episode.
4. Subjects entering the study must score at least 4 on the Clinical Global Impression Scale.
5. At least two weeks of ongoing treatment with current antipsychotic agents during the pre-treatment stabilization period.
6. Stable symptoms throughout the 2-week pre-treatment stabilization period. Clinical stability is defined as two consecutive weekly CGI ratings with no change in score, and with no more than a 20% change in PANSS total score.
7. No change in anticholinergic, benzodiazepine, or mood stabilizer medications for the pre-treatment stabilization period.
8. No anticipated need to alter any of the above medications (antipsychotics, anticholinergics, benzodiazepines, or mood stabilizers) for the 8-week duration of the study.
9. Ability to participate fully in the informed consent process, or have a legal guardian able to participate in the informed consent process.

Exclusion Criteria:

1. Evidence of serious neurologic or endocrine disorder, for example severe head trauma, seizure disorder, dementia, Cushings disease, or thyroid disorder, mental retardation, alcohol or drug abuse, substance dependence (other than nicotine dependence), or presenting symptoms likely substance-induced, as judged by a study physician.
2. Unstable medical illness or neurologic illness (seizures, CVA); history of prostate, breast, uterine, or ovarian cancer.
3. Pregnant women, use of oral contraceptives or other hormonal supplementation such as estrogen.
4. Current active suicidal and/or homicidal ideation, intent, or plan.
5. Known allergy to study medication.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The Clinical Global Impression Scale (CGI-S) The Positive and Negative Syndrome Scale (PANSS) The Scale for the Assessment of Negative Symptoms (SANS) | baseline, 2, 4, 6, and 8 weeks

SECONDARY OUTCOMES:
Global Assessment of Functioning | baseline, 2, 4, 6, and 8 weeks
The Cambridge Neuropsychological Test Automated Battery (CANTAB) | baseline, 4 and 8 weeks
Extrapyramidal Symptom Rating Scale | baseline, 2, 4, 6, and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Ritsher, MD, PhD, Study Chair — Technion and Shaar Menashe MHC; Anatoly Kreinin, MD, PhD, Study Director — Technion and Tirat Carmel Mental Health Center
Locations (1):
- Shaar Menashe MHC and Tirat Carmel MHC, Hadera, Israel

REFERENCES:
- [Background] Ritsner M, Maayan R, Gibel A, Weizman A. Differences in blood pregnenolone and dehydroepiandrosterone levels between schizophrenia patients and healthy subjects. Eur Neuropsychopharmacol. 2007 Apr;17(5):358-65. doi: 10.1016/j.euroneuro.2006.10.001. Epub 2006 Nov 21. PMID 17123790